CLINICAL TRIAL: NCT03133091
Title: Epidural Analgesia During Labour Randomized Clinical Trial Comparing Patient Controlled Epidural Analgesia Versus Patient Intermittent Epidural Boluses With Levobupivacaine
Brief Title: Epidural Analgesia During Labour
Acronym: PIEBvsPCEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, MARIA BELEN RODRIGUEZ-CAMPOO, PhD title in Medicine and Surgery, Hospital del Rio Hortega
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 290587
Record Dates: First submitted 2016-09-12; First posted 2017-04-28 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia, Obstetrical; Analgesia, Epidural
Keywords: PIEB; PCEA; LEVOBUPIVACAINE
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PIEB (Patient Intermittent Epidural Bolus) (Active Comparator): PIEB: The boluses are programmed every 30 minutes. The patient can ask for another extra bolus in between if she wishes.
  The dosis per hour are equivalent to the PCEA. We make a comparison between PCEA vs PIEB.
  Interventions: Drug: PIEB: Patient Intermittent Epidural Boluses
- PCEA (Patient continuous Epidural Analgesia) (Active Comparator): PCEA: There is a continuous infusion and the patient can order extra boluses every 15 minutes.
  The dosis per hour are equivalent to the other arm to the PIEB. We make a comparison between PCEA vs PIEB.
  Interventions: Drug: PCEA: Patient Controlled Epidural Analgesia

INTERVENTIONS:
Drug: PIEB: Patient Intermittent Epidural Boluses — Each patient were randomized to PIEB (7 ml bolus every 30 minutes, with extra boluses (PCEA) of 6 ml every 20 minutes) or PCEA (5 ml in continuous perfussion + PCEA of 5 ml every 15 minutes).
  Arms: PIEB (Patient Intermittent Epidural Bolus)
Drug: PCEA: Patient Controlled Epidural Analgesia — Each patient were randomized to PIEB (7 ml bolus every 30 minutes, with extra boluses (PCEA) of 6 ml every 20 minutes) or PCEA (5 ml in continuous perfussion + PCEA of 5 ml every 15 minutes).
  Arms: PCEA (Patient continuous Epidural Analgesia)

SUMMARY:
Randomized single blind trial based on comparing the way the local anesthetic is dosificated during labour. The pain control is evaluated and compared with both dosage techniques (PCEA vs PIEB)using levobupivacaine and fentanyl. The primary objective is to see no differences in pain control(VAS, Visual Analog Scale). The secondary goals are the differences in motor block(Bromage Scale), satisfaction (Likert Scale), the outcome (eutocic, instrumental o cesarean section), second stage of labour time, newborn´s Apgar and pH and total dosis and secondary effects of local anesthetic.

DETAILED DESCRIPTION:
There is a protocol where every healthy primiparous women have the chance to join the study after the explanation and the informed consent is signed. There are blind envelopes with the two kinds of treatment and the investigator only has to follow the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 20- 40 years-old women
* Primiparous women
* Dilatation 3- 7 cm
* No risk illnesses for epidural block
* No risk pregnancy
* Signed informed consent

Exclusion Criteria:

* Illnesses which are a risk for pregnancy
* Multiparous women
* Contraindicated diseases for epidural block
* Women who can not understand the procedure
* Women who do not want to sign the informed consent
* Patients with drug´s allergy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
VAS | 4 times after epidural block: previous, 1 hour after, 2 hours after, 15 minutes after delivery
  Change from baseline in Visual Analog Scale

SECONDARY OUTCOMES:
Satisfaction (Likert Scale) | 1 hour after delivery
  1 (very satisfied), 2 (satisfied), 3 (no comments), 4 (not very satisfied), 5 (not satisfied at all)
Bromage Scale | 15 minutes after Epidural Block and 1 hour after epidural block
Labour Outcome | Delivery
  Eutocic
Labour Outcome | Delivery
  instrumental
Labour Outcome | Delivery
  cesarean section
Expulsive time | From 10 cm of dilatation until delivery
Apgar at birth | 1 minute after birth
  Apgar measured in 1 minute
Apgar at birth | 5 minutes after birth
  Apgar measured in 5 minutes
fetal pH at birth | 0 minutes after delivery
  0 minutes after delivery
Total Dosis of Levobupivacaine | 0 minutes after delivery
  miligrams

CONTACTS AND LOCATIONS:
Overall Officials: M BELEN RODRIGUEZ-CAMPOO, Study Director — Resident
Locations (1):
- Hospital Universitario Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Result] Wong CA, Ratliff JT, Sullivan JT, Scavone BM, Toledo P, McCarthy RJ. A randomized comparison of programmed intermittent epidural bolus with continuous epidural infusion for labor analgesia. Anesth Analg. 2006 Mar;102(3):904-9. doi: 10.1213/01.ane.0000197778.57615.1a. PMID 16492849
- [Result] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Result] Chua SM, Sia AT. Automated intermittent epidural boluses improve analgesia induced by intrathecal fentanyl during labour. Can J Anaesth. 2004 Jun-Jul;51(6):581-5. doi: 10.1007/BF03018402. PMID 15197122
- [Result] Lin Y, Li Q, Liu J, Yang R, Liu J. Comparison of continuous epidural infusion and programmed intermittent epidural bolus in labor analgesia. Ther Clin Risk Manag. 2016 Jul 14;12:1107-12. doi: 10.2147/TCRM.S106021. eCollection 2016. PMID 27471390
- [Result] Halpern SH, Carvalho B. Patient-controlled epidural analgesia for labor. Anesth Analg. 2009 Mar;108(3):921-8. doi: 10.1213/ane.0b013e3181951a7f. PMID 19224805
- [Result] Gizzo S, Noventa M, Fagherazzi S, Lamparelli L, Ancona E, Di Gangi S, Saccardi C, D'Antona D, Nardelli GB. Update on best available options in obstetrics anaesthesia: perinatal outcomes, side effects and maternal satisfaction. Fifteen years systematic literature review. Arch Gynecol Obstet. 2014 Jul;290(1):21-34. doi: 10.1007/s00404-014-3212-x. PMID 24659334
- [Result] Melzack R. The myth of painless childbirth (the John J. Bonica lecture). Pain. 1984 Aug;19(4):321-337. doi: 10.1016/0304-3959(84)90079-4. No abstract available. PMID 6384895
- [Result] Hiltunen P, Raudaskoski T, Ebeling H, Moilanen I. Does pain relief during delivery decrease the risk of postnatal depression? Acta Obstet Gynecol Scand. 2004 Mar;83(3):257-61. doi: 10.1111/j.0001-6349.2004.0302.x. PMID 14995921
- [Result] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Result] Eriksen LM, Nohr EA, Kjaergaard H. Mode of delivery after epidural analgesia in a cohort of low-risk nulliparas. Birth. 2011 Dec;38(4):317-26. doi: 10.1111/j.1523-536X.2011.00486.x. Epub 2011 Sep 6. PMID 22112332
- [Result] Lieberman E, Lang JM, Cohen A, D'Agostino R Jr, Datta S, Frigoletto FD Jr. Association of epidural analgesia with cesarean delivery in nulliparas. Obstet Gynecol. 1996 Dec;88(6):993-1000. doi: 10.1016/s0029-7844(96)00359-6. PMID 8942841
- [Result] Patel RR, Peters TJ, Murphy DJ; ALSPAC Study Team. Prenatal risk factors for Caesarean section. Analyses of the ALSPAC cohort of 12,944 women in England. Int J Epidemiol. 2005 Apr;34(2):353-67. doi: 10.1093/ije/dyh401. Epub 2005 Jan 19. PMID 15659468
- [Result] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Derived] Rodriguez-Campoo MB, Curto A, Gonzalez M, Aldecoa C. Patient intermittent epidural boluses (PIEB) plus very low continuous epidural infusion (CEI) versus patient-controlled epidural analgesia (PCEA) plus continuous epidural infusion (CEI) in primiparous labour: a randomized trial. J Clin Monit Comput. 2019 Oct;33(5):879-885. doi: 10.1007/s10877-018-0229-x. Epub 2018 Nov 30. PMID 30506299